CLINICAL TRIAL: NCT03097367
Title: Predictor of Early Recovery on Urinary Continence After Laparoscopic Radical Prostatectomy: Bladder Neck Level and the Association With Urodynamic Parameters
Brief Title: Predictor of Early Recovery on Urinary Continence After Laparoscopic Radical Prostatectomy
Status: Completed | Type: Observational
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Hann-Chorng Kuo, Chaiman, Department of Urology, Buddhist Tzu Chi General Hospital
Other Study IDs: TCGH106-42-B
Record Dates: First submitted 2017-03-27; First posted 2017-03-31 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Urinary Incontinence
Keywords: laparoscopic radical prostatectomy; urinary incontinence; prostate cancer; bladder neck level; urodynamics
MeSH Terms: conditions — Urinary Incontinence; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: bladder neck level on cystography — All patients had investigated by retrograde cystography after LRP and were grouped according their bladder neck position: Level 0: bladder neck at or above the superior margin of the symphysis pubis (SMSP), Level -1: bladder neck at <2 cm below SMSP, and Level -2: bladder neck at >2 cm below SMSP.
  Other Names: BN level

SUMMARY:
To investigate the relationship between post-operative bladder neck levels and urodynamic parameters and their effect on urinary incontinence after laparoscopic radical prostatectomy (LRP). Forty-eight consecutive patients undergoing LRP were retrospectively reviewed. All patients had investigated by retrograde cystography after LRP and were grouped according their bladder neck position: Level 0: bladder neck at or above the superior margin of the symphysis pubis (SMSP), Level -1: bladder neck at <2 cm below SMSP, and Level -2: bladder neck at >2 cm below SMSP. Urodynamic studies were carried out at baseline, 3 and 6 months post-operatively. Early recovery of urinary continence was defined as no urine leakage or only one pad/day used within 3 months after surgery. Demographic characteristics, changes of urodynamic parameters and continence outcomes were analyzed.

DETAILED DESCRIPTION:
Laparoscopic radical prostatectomy (LRP) is effective in treating localized prostate cancer with good long-term oncological outcomes. Urinary incontinence, which is a bothersome complication with a negative effect on the patient's quality of life, remains a relevant problem after LRP, despite the improvements in the surgical technique. More than 80% of patients undergoing radical prostatectomy encounter urinary incontinence immediately after catheter removal, but the bladder condition can generally stabilize within two years after operation. Among the patients undergoing LRP, persistent urinary incontinence has been reported in 4-30% of patients, and further treatment is often required.

Definite evaluation for the voiding function has been recommended for patients with prolonged post-prostatectomy urinary incontinence (PPI). To improve quality of life after LRP, early recovery of urinary continence is an important concern for patients. Several studies have investigated the predictive factors of early recovery of urinary continence after prostatectomy, including the amount of urine loss after catheter removal, pelvic floor muscle function, a nerve-sparing technique, and the membranous urethral length loss ratio.

Other factors relating to the early recovery of urinary continence include post-operative anatomy of the lower urinary tract, such as the length of the membranous urethra and the level of the vesicourethral junction. However, there has been no consensus on the standard criteria that should be used to measure the structural changes, and the relationship between the urodynamic change and the anatomical morphology remains unclear. In this study, investigators study the relationship between the urodynamic parameters and the bladder neck levels after LRP, and their effects on the early recovery of urinary incontinence.

This study was a retrospective analysis. From 2011 to 2014, a total of 48 consecutive patients with localized prostatic cancer underwent LRP in single medical center by two experienced surgeons. Videourodynamic study was performed before operation (baseline) and at 3 and 6 months after operation. The Ethics Committee of the hospital approved this study and written informed consent was waived because the study was a retrospective analysis. The principles of Helsinki Declaration were followed throughout the study.

The urodynamic parameters were measured and recorded including first sensation of filling (FSF), maximum flow rate (Qmax), detrusor pressure at Qmax (PdetQmax), voided volume, cystometric bladder capacity (CBC), bladder compliance, post-void residual (PVR) volume, maximal urethral closure pressure (MUCP) and functional profile length (FPL). The urodynamic parameters were compared between baseline and different time-points after LRP.

The BN level was evaluated by retrograde cystography, which was routinely performed 7 to 14 days after LRP to evaluate the condition of anastomosis. The image was obtained anteroposteriorly after infusing 100-150 mL of contrast solution into the bladder while the patient was in standing position. The distance between the bladder neck and the superior margin of the symphysis pubis (SMSP) was then measured by the same urologist. The bladder neck level was graded on a three-point scale: a bladder neck level at or above the SMSP was marked as level 0, a bladder neck level with a distance less than 2 cm below the SMSP was marked as level -1, and bladder neck levels 2 or more cm below the SMSP was labeled as level -2.

The patient's urinary continence status was evaluated on direct visits and via questionnaires during follow-up periods at 3, 6, and 12 months post-operatively. Patients without urine leakage in their daily life and those who used only one pad per day for safety reasons without limitation in their daily activities were defined as "urinary continent". Otherwise, the patients were defined as "urinary incontinent". Regaining continence within 3 months after LRP was considered early recovery of urinary continence.

The data was collected retrospectively by chart review. The variables among continent and incontinent patients were evaluated by univariate analysis (t-test for continuous variables and Chi-square for categorical variables ). The ANOVA test was use to compare the urodynamic parameters between different BN levels. Statistical analysis was performed using SPSS 20.0 statistical software.

ELIGIBILITY:
Inclusion Criteria:

* Patients with localized prostate cancer underwent laparoscopic radical prostatectomy

Exclusion Criteria:

* Patients who did not have regular follow-up after surgery

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with localized prostate cancer underwent laparoscopic radical prostatectomy
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
urinary continence at 3 months after laparoscopic radical prostatectomy | from baseline to 3 months
  Patients without urine leakage in their daily life and those who used only one pad per day for safety reasons without limitation in their daily activities at 3 months after laparoscopic radical prostatectomy were defined as "urinary continent"

CONTACTS AND LOCATIONS:
Overall Officials: HannChorng Kuo, M.D., Principal Investigator — Buddhist Tzu Chi General Hospital

IPD SHARING:
Plan to Share IPD: No
No plan to share data with other researchers